CLINICAL TRIAL: NCT05649761
Title: A Phase I, Open-label, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of QL1604, a Humanized Anti-PD-1 Monoclonal Antibody, in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study of QL1604 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1604-001
Record Dates: First submitted 2022-11-24; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1604 injection (Experimental): Participants will receive QL1604 injection 0.3 mg/kg,1mg/kg, 3mg/kg,10mg/kg, or 200mg intravenous every 2 weeks or every 3 weeks and will be continued until disease progression or unacceptable toxicity.
  Interventions: Drug: QL1604 injection

INTERVENTIONS:
Drug: QL1604 injection — Participants will receive QL1604 injection 0.3 mg/kg,1mg/kg, 3mg/kg,10mg/kg, or 200mg intravenous every 2 weeks or every 3 weeks and will be continued until disease progression or unacceptable toxicity.

SUMMARY:
This is a first-in-human (FIH), dose-escalation, PK expansion, monotherapy efficacy expansion, and open-label phase I clinical study assessing the safety, tolerability, pharmacokinetics, immunogenicity, and preliminary efficacy of QL1604 injection （a humanized anti-PD-1 monoclonal antibody）in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this clinical study; completely understand and know this study as well as sign the informed consent form (ICF);
2. Age ≥ 18 years and ≤ 70 years when ICF is signed;
3. Pts with histologically or cytologically confirmed advanced solid tumors;
4. At least one target lesion as defined per RECIST Version (v) 1.1;
5. Subjects who have disease progression or intolerable reactions after the currently available standard anti-cancer treatment previously received or refused prior cancer therapy regimen(s) ;
6. Eastern Cooperative Oncology Group performance status of 0 or 1;
7. Life expectancy of greater than 12 weeks;
8. Adequate hematologic and organ function;
9. Female subjects who are not pregnant or breastfeeding
10. Male and female subjects able to have children must agree to use highly effective method of contraception throughout the study and for at least 120 days after last dose;

Exclusion Criteria:

1. Known hypersensitivity to any monoclonal antibody, QL1604 and/or any of its excipients;
2. Active autoimmune disease that has required systemic treatment, replacement therapy is acceptable;
3. Subjects with major cardiovascular and cerebrovascular diseases;
4. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of study drug;
5. Subjects who have received surgery, radiotherapy, chemotherapy, targeted therapy, other anti-tumor treatments, or participating in other clinical studies is less than 4 weeks before the first administration of investigational product;
6. Received a live vaccine;
7. Infection with human immunodeficiency virus (HIV);
8. Known psychiatric or substance abuse disorders that would interfere with the requirements of the study;
9. History or current evidence of any condition, therapy, or laboratory abnormality, that might confound the results of the trial, or interfere with the participant's participation for the full duration of the study, or investigators/sponsor consider the subjects are not suitable for this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2023-01-23 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 21 days after the first dose
  Dose-limiting toxicity (DLT)
maximum tolerated dose(MTD) | Up to 21 days after the first dose
  maximum tolerated dose(MTD)
recommended phase II dose (RP2D) | up to 2 years
  recommended phase II dose (RP2D)

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment-Related AEs | up to 2 years
  according to NCI CTCAE V5.0
Maximum Concentration (Cmax) of QL1604 in Solid Tumor Participants | up to 2 years
  Maximum Concentration (Cmax)
Time to Maximum Concentration (Tmax) of QL1604 in Solid Tumor Participants | up to 2 years
  Time to Maximum Concentration (Tmax)
Terminal Half-Life (t ½) of QL1604 in Solid Tumor Participants | up to 2 years
  Terminal Half-Life (t ½)
Area Under the Concentration-Time Curve of QL1604 From Time 0 to Day 28 (AUC 0-22) in Solid Tumor Participants | up to 22 days
  Area Under the Concentration-Time Curve
Objective Response Rate (ORR) According to RECIST 1.1 | up to 2 years
  Objective Response Rate (ORR) According to RECIST 1.1
Disease Control Rate (DCR) According to RECIST 1.1 | up to 2 years
  Disease Control Rate (DCR) According to RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of The University of Chinese Academy of Sciences, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Z, Xu Y, Hong W, Gong L, Chen K, Qin J, Xie F, Wang F, Tian X, Meng X, Feng W, Li L, Zhang B, Kang X, Fan Y. A first-in-human, open-label, dose-escalation and dose-expansion phase I study to evaluate the safety, tolerability, pharmacokinetics/pharmacodynamics, and antitumor activity of QL1604, a humanized anti-PD-1 mAb, in patients with advanced or metastatic solid tumors. Front Immunol. 2023 Oct 23;14:1258573. doi: 10.3389/fimmu.2023.1258573. eCollection 2023. PMID 37936687